CLINICAL TRIAL: NCT02600182
Title: Effects of Bilevel Positive Airway Pressure in Postoperative Cardiac Surgery: A Randomized Clinical Trial
Brief Title: Bilevel Positive Airway Pressure in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Antônio Marcos Vargas da Silva (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Antônio Marcos Vargas da Silva, PhD in Physiology, Universidade Federal de Santa Maria
Organization: Universidade Federal de Santa Maria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDAAA 801
Record Dates: First submitted 2015-11-02; First posted 2015-11-09 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Cardiopathy; Surgery
Keywords: Thoracic surgery; Non-invasive ventilation; Physiotherapy
MeSH Terms: conditions — Heart Diseases | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilevel Positive Airway Pressure (BiPAP) (Experimental): The routine physical therapy will be performed in two groups (control and BiPAP). The BiPAP group will receive two daily sessions of 20 minutes, with positive expiratory pressure of 10cmH2O and inspiratory of 15cmH2O.
  Interventions: Device: Bilevel Positive Airway Pressure
- Control (No Intervention): Routine physical therapy will be performed.

INTERVENTIONS:
Device: Bilevel Positive Airway Pressure — Bilevel positive airway pressure twice per day during the hospital stay.
  Other Names: BiPAP
  Arms: Bilevel Positive Airway Pressure (BiPAP)

SUMMARY:
The purpose of this study was to determine the effects of Bilevel Positive Airway Pressure (BiPAP) on variables clinics, cardiorespiratory and physical functional in patients undergoing cardiac surgery at the University Hospital of Santa Maria.

DETAILED DESCRIPTION:
This randomized controlled trial aimed to evaluate the effects of Bilevel Positive Airway Pressure (BiPAP) in patients undergoing heart surgery of valve replacement and coronary artery bypass graft on the variables clinics, cardiorespiratory and physical functional.These individuals were randomized to compose the control group (GC) and the BiPAP group (GBiPAP). The routine physical therapy was performed in both groups and in the BiPAPG two daily sessions of 20 minutes were applied with positive expiratory pressure of 10cmH2O and inspiratory of 15cmH2O. To verify the effect of this intervention, before and after the protocol patients underwent the following evaluations: the 6-minute walk test (6MWT), the heart rate variability, the manovacuometry, and cirtometry in the axillary line, umbilical line and the xiphoid appendix.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients in preoperative for coronary artery bypass or valve replacement.

Exclusion Criteria:

* Inability to understand or sign a free and informed consent form
* Chronic obstructive pulmonary disease (COPD)
* Cerebrovascular disease
* Musculoskeletal disease
* Chronic infectious disease
* Unstable angina
* Treatment with steroids, hormones or chemotherapy for cancer
* Prolonged mechanical ventilation
* Unable of maintaining airway patency
* Severe hemodynamic instability
* Abdominal distension or vomiting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Peripheral Oxygen Saturation by pulse oximetry | up to 36 weeks

SECONDARY OUTCOMES:
Vital Signs | up to 36 weeks
Length of stay | up to 36 weeks
Postoperative complications | up to 36 weeks
Six-minute walk test (6MWT) | up to 36 weeks
Heart rate variability by a pulse frequency meter | up to 36 weeks
Maximum inspiratory pressure by a digital pressure transducer (manovacuometry) | up to 36 weeks
Maximum expiratory pressure by a digital pressure transducer (manovacuometry) | up to 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antônio M Vargas da Silva, PhD, Principal Investigator — Universidade Federal de Santa Maria
Locations (1):
- Federal University of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided